CLINICAL TRIAL: NCT05544526
Title: Chimeric Antigen Receptor (CAR)-T Cells to Target GD2 for Diffuse Midline Glioma
Brief Title: CAR T Cells to Target GD2 for DMG
Acronym: CARMIGO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/ 150853
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: CAR T cells; Diffuse Midline Glioma; DMG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GD2 CAR T Cells (Experimental): Treatment with the ATIMP: GD2 CAR T-cells
  Interventions: Biological: GD2 CAR T cells

INTERVENTIONS:
Biological: GD2 CAR T cells — Infusion with: GD2 CAR T-cells

SUMMARY:
The CARMIGO Trial is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in children and young adults aged 2-16 years with Diffuse Midline Glioma (DMG).

The study will evaluate the feasibility of generating the ATIMP, the safety and tolerability of the GD2CAR T-cell therapy and how effectively GD2CAR T-cells engraft, expand and persist following administration in patients with DMG.

DETAILED DESCRIPTION:
The CARMIGO Trial is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in children and young adults aged 2-16 years with Diffuse Midline Glioma (DMG).

The ATIMP for this study is cryopreserved autologous patient-derived T-cells transduced with GD2CAR vector to generate GD2CAR T-cells.

Patients will undergo an unstimulated leucapheresis for the generation of the ATIMP which will take approximately 15 days to generate.

Patients will have an intraventricular catheter (Ommaya catheter) placed following enrolment and prior to GD2 CAR T cell infusion to allow monitoring, and treatment if necessary, of increased intracranial pressure (ICP).

Patients will receive lymphodepleting (LD) chemotherapy with fludarabine 30mg/m2 administered over 4 days (Day -6 to Day -3) and cyclophosphamide 60mg/kg administered over 2 days (Day -4 and Day-3).

All patients will be treated on Theme 1 of the study (intravenous CAR T administration) at one of the three dose levels (Dose Level 1: 3 x10^7 GD2 CAR T cells/m2; Dose Level 2: 10 x10^7 GD2 CAR T cells/m2; Dose Level 3: 30 x10^7 GD2 CAR T cells/m2) following LD chemotherapy as described above. Patients with no/partial response at Day 28 (or disease progression after initial CR beyond Day 28) and in the absence of severe/persisting toxicity related to the ATIMP, will be potentially eligible for Theme 2 of the study where they can receive Dose 2, a single dose of 30 x 10^6 CD19CAR T-cells intraventricularly via an Ommaya reservoir following LD chemotherapy as described above.

The study will evaluate the feasibility of generating the ATIMP, the safety of administering GD2CAR T-cell therapy, the tolerability of the GD2CAR T cell in patients and how effectively GD2CAR T-cells engraft, expand and persist following administration in patients with DMG.

Following infusion of GD2CAR T-cell therapy patients will be monitored for between 2-4 weeks as an inpatient. Following discharge, patients will enter the interventional follow up phase and be followed up for 1 year. Patients will be seen at 6 weeks post infusion then 3 monthly until 1 year post GD2CAR T-cell infusion.

If patients relapse within the first year post last GD2CAR T-cell infusion they will come off the interventional follow up and will be followed up annually until the end of trial is declared.

After completing the 1 year interventional phase of the study all patients, irrespective of whether they progressed or responded to treatment, will enter long term follow up until the end of trial is declared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 and ≤ 16 years
2. Tissue diagnosis of H3K27M mutant Diffuse Midline Glioma.
3. Radiographically evident tumour restricted to the brain stem or spinal cord.
4. At least 6 weeks following completion of radiation therapy.
5. At least 3 weeks or 5 half-lives, whichever is shorter, after treatment with agents on other early phase clinical trial
6. Performance status: Karnofsky (age ≥ 10 years) or Lansky (age < 10) score ≥ 40% allowing for stable neurological deficit due to DMG
7. Absolute neutrophil count ≥1.5 x109/L and platelet count ≥ 100 x109/L
8. Total bilirubin < 1.5 ULN and ALT < 2.5 ULN
9. Serum creatine < 1.5 ULN for age.
10. For post-pubertal subjects agreement to have a pregnancy test, use adequate contraception (if applicable)
11. Written informed consent

Exclusion Criteria:

1. Systemic corticosteroid therapy ≥ 0.05 mg/kg dexamethasone daily (or equivalent) at time of RQR8/huK28Z CAR T cell infusion
2. Tumour involvement of the thalamus or supratentorial lesions, cerebellar vermis or hemispheres (pontocerebellar peduncle involvement is allowed)
3. Clinical or radiological evidence of true tumour progression
4. Active hepatitis B, C or HIV infection
5. Inability to tolerate leukapheresis
6. Pre-existing significant neurological disorder not related to DMG
7. Clinically significant systemic illness or medical condition (e.g., significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgement of the investigator is likely to interfere with assessment of safety or efficacy of the investigational regimen and its requirements.
8. Any contraindication to lymphodepletion or to the use of Cyclophosphamide or Fludarabine as per the local SmPC
9. Any contraindication to the use of Anticoagulant Citrate Dextrose Solution
10. Any contraindication to Ommaya reservoir insertion (or similar catheter)
11. Known allergy to albumin, DMSO or EDTA
12. Primary immunodeficiency or history of autoimmune disease (e.g., Crohn's, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression /systemic disease modifying agents within the last 2 years
13. Prior treatment with investigational or approved gene therapy or cell therapy products
14. Life expectancy <3 months
15. Use of rituximab (or rituximab biosimilar) within the last 3 months prior to RQR8/huK28Z CAR T cell infusion
16. Post-pubertal subjects who are pregnant or breastfeeding

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP | 28 days
  Toxicity of GD2 CAR T cells as assessed by the incidence of grade 3-5 toxicity causally related to the ATIMP (particularly severe cytokine release syndrome and severe neurotoxicity).
Feasibility of manufacturing GD2 CAR T-cells evaluated by the number of therapeutic products generated | 28 days
  Feasibility of generation of the ATIMP as evaluated by the number of therapeutic products generated and the number of ATIMPs infused (as an intravenous agent (Theme 1) and as an intraventricular agent (Theme 2) after successful manufacture.

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  The proportion of patients alive at 1 year will be tabulated. If numbers are sufficient, overall survival will also be analysed using Kaplan-Meier survival analyses. Survival times will be measured from the date of GD2 CAR T infusion until the date of death from any cause.
Progression Free Survival (PFS) | 1 year
  The proportion of patients alive and progression-free at 1 year will be tabulated. Progression-free survival will be analysed using Kaplan-Meier survival analyses with the median survival time reported. Survival times will be measured from the date of the GD2 CAR T infusion until the date of progression or death.
Time to Progression (TTP) | 1 year
  TTP will be summarised as a median and range. If numbers are sufficient, this will also be analysed using Kaplan-Meier survival analyses with the duration calculated as the time from first response (≥PR) until progression
Best objective response rate (ORR) | 1 year
  This will be taken as the best response as defined by RAPNO criteria observed at any time point following CAR T infusion. The number and proportion of patients achieving a response ≥PR will be presented for all patients as well as by dose level.

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No